CLINICAL TRIAL: NCT00133744
Title: Impact of Iron/Folic Acid Versus Multimicronutrient Versus Folic Acid Supplements During Pregnancy on Mortality, Morbidity, and Complications During Pregnancy, Labor, and Delivery: A Randomized Controlled Trial in China
Brief Title: Impact of Prenatal Vitamin/Mineral Supplements on Perinatal Mortality
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Zuguo Mei, Ceanters for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-4084
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Perinatal Mortality; Stillbirth; Neonatal Mortality
Keywords: pregnancy; vitamins; minerals; supplements; mortality; prenatal; perinatal; anemia; birthweight; preterm; iron; micronutrients; Stillbirths; Early neonatal deaths
MeSH Terms: conditions — Perinatal Death; Stillbirth; Anemia; Birth Weight; Premature Birth | interventions — Folic Acid; Iron; Geritol; Minerals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A, 1 (Active Comparator)
  Interventions: Dietary Supplement: folic acid
- A, 2 (Experimental)
  Interventions: Dietary Supplement: folic acid plus iron
- A, 3 (Experimental): Multiple micronutrient supplement
  Interventions: Dietary Supplement: supplements with multiple vitamins and minerals

INTERVENTIONS:
Dietary Supplement: folic acid — pills by mouth, one per day, from the first prenatal visit until delivery, 400 micrograms (mcg) folic acid
  Arms: A, 1
Dietary Supplement: folic acid plus iron — pills by mouth, one per day, from the first prenatal visit until delivery, 400 mcg folic acid, 30 mg Fe
  Arms: A, 2
Dietary Supplement: supplements with multiple vitamins and minerals — pills, one per day, from the first prenatal visit until delivery; folic acid 400 mcg, Fe 30 mg, vitamin(vit) A 800 mcg, vit E 10 mg, vit D 5 mcg, vit C 70 mg, vit B1 1.4 mg, vit B2 1.4 mg, vit B6 1.9 mg, vit B12 2.6 mcg, Niacin 18 mg, Zn 15 mg, Cu 2mg, Iodine 150 mcg, Selenium 65 mcg
  Other Names: UNIMMAP
  Arms: A, 3

SUMMARY:
The purpose of this study is to determine whether a daily prenatal supplement of iron plus folic acid or a daily prenatal supplement with multiple vitamins and minerals given to women from their first prenatal visit through delivery reduces perinatal mortality compared with a daily prenatal supplement of folic acid alone.

DETAILED DESCRIPTION:
In the project area in China, the rate of perinatal mortality (stillbirths and infant deaths within 6 days of birth) is two times that of the United States. Causes of perinatal mortality include, but are not limited to, low birth weight and preterm delivery. Anemia (low hemoglobin) among pregnant women is associated with low birth weight and preterm delivery and also is elevated in the project area. Supplements of iron, folic acid, and other vitamins and minerals can prevent anemia among pregnant women, but the effects of these supplements on other maternal and infant health outcomes are unclear.

Since 1993, the People's Republic of China has recommended that newly married women, and those who plan pregnancy, take 400μg of folic acid daily through the first trimester of pregnancy. Although WHO recommends that pregnant women take iron and folic acid supplements, there is currently no national recommendation that pregnant women in China take iron or other vitamin or mineral supplements (other than folic acid). UNICEF is now testing a prenatal vitamin and mineral supplement in programs to prevent low birth weight. Our study will provide additional information about the health impact of the UNICEF prenatal supplement versus an iron and folic acid supplement versus folic acid alone.

Comparisons:

* Infants of women who receive daily prenatal supplements that contain 400μg folic acid alone, will be compared with infants of women who receive daily supplements that contain 30 mg iron and 400 μg folic acid.
* Infants of women who receive daily supplements that contain 30 mg iron and 400 μg folic acid will be compared with infants of women who receive a daily supplement containing 30 mg iron, 400μg folic acid and other vitamins and minerals (UNICEF formulation).

ELIGIBILITY:
Inclusion Criteria:

* Live in one of the study counties (Laoting, Mancheng, Fengrun, Xianghe, Yuanshi)
* Can follow instructions
* Can swallow pills

Exclusion Criteria:

* >= 20 weeks gestation at enrollment
* Previous live birth
* Anemic (hemoglobin [Hb] <10 g/dl in 1st trimester and < 9.5 g/dl in 2nd trimester) at enrollment
* Current use of iron or other vitamin or mineral supplements (except folic acid)
* Age < 20 years at enrollment
* Under treatment for anemia at enrollment
* Refuse to participate

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18962 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Perinatal mortality, i.e., the number of stillbirths (fetal deaths of 28 weeks or more of gestation) and the number of deaths within the first 0-6 days of life per 1000 births (live births and stillbirths) | 20 weeks gestation to 6 days postpartum

SECONDARY OUTCOMES:
Maternal anemia | 24-28 weeks gestation
Maternal anemia | 4-8 weeks postpartum
Infant gestational age at birth, preterm delivery | delivery
Infant birth weight, low birth weight | at birth
Infant low weight-for-height | infant age 6 months and 12 months
Infant anemia | 6 months and 12 months of age
maternal gastrointestinal side effects | monthly from a month after enrollment until delivery

CONTACTS AND LOCATIONS:
Overall Officials: Weicheng You, MD, MBA, Principal Investigator — Peking University Health Science Center, Beijing China; Jianmeng Liu, MD, PhD, Study Director — Institute of Reproductive and Child Health, Peking University Health Science Center, Beijing China
Locations (5):
- China (5):
  - Fengrun Maternal and Child Health Institute, Fengrun, Hebei
  - Yuanshi Maternal and Child Health Institute, Huaiyang, Hebei
  - Laoting Maternal and Child Health Institute, Laoting, Hebei
  - Mancheng Maternal and Child Health Institute, Mancheng, Hebei
  - Xianghe Maternal and Child Health Institute, Xianghe, Hebei

REFERENCES:
- [Derived] Si KY, Li HT, Zhou YB, Li ZW, Zhang L, Zhang YL, Ye RW, Liu JM. Cesarean delivery on maternal request and common child health outcomes: A prospective cohort study in China. J Glob Health. 2022 Feb 26;12:11001. doi: 10.7189/jogh.12.11001. eCollection 2022. PMID 35265334
- [Derived] Liu Y, Li N, Mei Z, Li Z, Ye R, Zhang L, Li H, Zhang Y, Liu JM, Serdula MK. Effects of prenatal micronutrients supplementation timing on pregnancy-induced hypertension: Secondary analysis of a double-blind randomized controlled trial. Matern Child Nutr. 2021 Jul;17(3):e13157. doi: 10.1111/mcn.13157. Epub 2021 Feb 16. PMID 33594802
- [Derived] Chen S, Li N, Mei Z, Ye R, Li Z, Liu J, Serdula MK. Micronutrient supplementation during pregnancy and the risk of pregnancy-induced hypertension: A randomized clinical trial. Clin Nutr. 2019 Feb;38(1):146-151. doi: 10.1016/j.clnu.2018.01.029. Epub 2018 Feb 15. PMID 29428785
- [Derived] Zhang Y, Jin L, Liu JM, Ye R, Ren A. Maternal Hemoglobin Concentration during Gestation and Risk of Anemia in Infancy: Secondary Analysis of a Randomized Controlled Trial. J Pediatr. 2016 Aug;175:106-110.e2. doi: 10.1016/j.jpeds.2016.05.011. Epub 2016 Jun 2. PMID 27263403
- [Derived] Liu JM, Mei Z, Ye R, Serdula MK, Ren A, Cogswell ME. Micronutrient supplementation and pregnancy outcomes: double-blind randomized controlled trial in China. JAMA Intern Med. 2013 Feb 25;173(4):276-82. doi: 10.1001/jamainternmed.2013.1632. PMID 23303315